CLINICAL TRIAL: NCT05723029
Title: Comparative Effects of Bowen Technique and Post Isometric Relaxation on Pain, Range of Motion and Hamstring Flexibility in Knee Osteoarthritis Patients
Brief Title: Bowen Technique and Post Isometric Relaxation in Knee Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0156
Record Dates: First submitted 2023-01-24; First posted 2023-02-10 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis
Keywords: Post Isometric Relaxation; Bowen Technique; Hamstring muscle flexibility; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Bowen Technique (Experimental): The subjects will receive Bowen Technique. The treatment session will be 3 times per week for 4 weeks for 20 minutes. The Bowen technique is a subtle and precise mobilization called Bowen moves. The mobilization is applied by using the fingers and thumbs over muscles, tendon, nerves and fascia. Only gentle non-invasive pressure is applied. A Bowen moves challenges the muscles for several seconds by the application of a gentle lateral pressure applied by the therapist thumb, against its medial edge. The muscle fibres and its fascia are disturbed from their neutral position and they are slightly stretched. The therapist apply gentle pressure towards the muscles using the skin slack available, and then rolls the thumb across the muscles and gently compressing it, the muscle will bounce back to its original position. The therapist has a sense of tissue tension, and this enables his/her to feel where stress has built up in the tissue.
  Interventions: Other: Bowen Technique
- Group B: Post Isometric Relaxation Technique (Experimental): The subjects will receive Post Isometric Relaxation Technique. Treatment session includes 3 times per week for 4 weeks for 20 minutes. Evaluation will be done before and after the treatment at the end of the 4th week. The outcome will be measured by the Active Knee Extension test, Numeric pain Rating Scale, and Goniometer. Post Isometric Relaxation is performed in supine position on treatment table. The therapist passively flexed the hip and knee at the 90 degrees and then passively extends the knee until the point of tissue resistance. Patient placed their leg on therapist shoulder and contracts his hamstring muscles by pushing down on the therapist shoulder for 10 seconds. After the contraction, patient is asked to relax, then therapist passively stretch to gain new range of muscles. The intervention is performed three times in a single session with 30 seconds rest intervals.
  Interventions: Other: Post Isometric Relaxation

INTERVENTIONS:
Other: Bowen Technique — A Bowen moves challenges the muscles for several seconds by the application of a gentle lateral pressure applied by the therapist thumb, against its medial edge. The muscle fibres and its fascia are disturbed from their neutral position and they are slightly stretched. The therapist apply gentle pressure towards the muscles using the skin slack available, and then rolls the thumb across the muscles and gently compressing it, the muscle will bounce back to its original position.
  Arms: Group A: Bowen Technique
Other: Post Isometric Relaxation — Post Isometric Relaxation is performed in supine position on treatment table. The therapist passively flexed the hip and knee at the 90 degrees and then passively extends the knee until the point of tissue resistance. Patient placed their leg on therapist shoulder and contracts his hamstring muscles by pushing down on the therapist shoulder for 10 seconds. After the contraction, patient is asked to relax, then therapist passively stretch to gain new range of muscles.
  Arms: Group B: Post Isometric Relaxation Technique

SUMMARY:
The Hamstring muscles are present at the posterior surface of the thigh. The muscles start in the gluteal region and run back of the thigh and insert into the popliteal fossa. The function of hamstring muscles flexes the knee and extension of the thigh. In degenerative joint disease, muscles tightness of the lower extremity leads to a decrease in joint flexibility. In knee joint osteoarthritis, hamstring muscles are more prone to tightness. The objective of this study is to compare the effects of the Bowen technique and Post Isometric Relaxation on pain, range of motion, and hamstring flexibility in knee osteoarthritis patients.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial and will be conducted at Al- Mustafa Medical and Physiotherapy Center. The study will be completed within the time duration of six months. For data collection, a convenient sampling technique will be used. The Population will be diagnosed with osteoarthritis patients. A sample size of total 24 patients will be taken in this study. The measurement tool will be Active knee extension test, Goniometer and Numeric pain rating scale. The pre-test and post-test outcome measurement will be taken. Patients will be divided into two groups. Group A will receive the Bowen technique intervention and Group B will receive the Post Isometric Relaxation technique. The interventions groups will receive three sessions per week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic subjects with hamstring tightness
* Both male and female
* Age between 45 to 65
* O degree to 20-degree active knee extension loss
* Subject with inter-articular knee joint pathology
* Diagnosed osteoarthritis patients
* Grade 1 to 4 Osteoarthritis

Exclusion Criteria:

* Subject history of lower extremity injury
* Any Neurological symptoms or radiating pain
* Any lower limb deformity
* Any fracture or Surgery is done for knee

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Active knee extension test | Baseline measurement (Pre-Treatment) in start on 1st day and post treatment follow-up for change will be taken on 4th week
  In this test, the subject is on the left-side lying on the examination table for bony landmark identification. The lateral femoral condyle, head of a fibula, and lateral malleolus of the right leg are marked to ensure that the same reference point is used for repeated measurement. When the landmarks are identified, the subject is instructed to lie in the supine position. The subject flexes the right hip at 90 degrees and grasps behind the right knee to stabilize the hip at 90 degrees. A goniometer is used to position the right knee at 90 degrees. A stationary arm long lateral femur and movable arm aligned with lateral fibula keeping lateral femoral condyle as an axis. The Patient actively extends the right knee as much as possible without moving the thigh from a vertical position. The active Range of motion of the knee is measured by a goniometer. (7) The active knee extension test have excellent intra-rater reliability(r = .7).
Change in Numeric pain rating scale | Baseline measurement (Pre-Treatment) in start at at 1st week and post treatment follow-up for change will be taken on4th week
  The Numeric pain rating scale is a self-reported measurement tool consisting of a numerical point scale. The scale is set up on a horizontal or vertical line, which ranges most commonly from 0 to 10, where 0 is no pain and 10 is the worst pain. The patient is asked to rate his or her pain intensity. There are three categories of pain least pain, average pain and, worst pain. The test-retest reliability for the Numeric pain rating scale varies from 0.67 to 0.96.
Change in Goniometer test | Baseline measurement (Pre-Treatment) in start on 1st day and post treatment follow-up for change will be taken on 4th week
  In this test, each subject is in the supine position, while a small pillow is placed beneath his head and neck. Then the legs and thighs of the other lower extremity are fixed to the bed with a strap. The knee flexion axis is being marked by a pen and from this point; a line is being drawn to the greater trochanter of the femur and one other line to the external malleolus of the ankle. These lines are used to measure the knee joint angles. The goniometer axis is placed on the knee axis and its arm is the place along with the line drawn on the thigh and the other arm is placed along with the line drawn on the leg. The Hip joint is 90 degrees and the vertical position of the thigh is being maintained. The subject is asked to do the active Knee extension slowly while the ankle is in the neutral position.

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, Mphil, Principal Investigator — Riphah International University
Locations (1):
- Al-Mustafa Medical and Physiotherapy Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahl C, Cleland JA. Visual analogue scale, numeric pain rating scale and the McGill Pain Questionnaire: an overview of psychometric properties. Physical therapy reviews. 2005;10(2):123-8.
- [Background] Shamsi M, Mirzaei M, Khabiri SS. Universal goniometer and electro-goniometer intra-examiner reliability in measuring the knee range of motion during active knee extension test in patients with chronic low back pain with short hamstring muscle. BMC Sports Sci Med Rehabil. 2019 Mar 22;11:4. doi: 10.1186/s13102-019-0116-x. eCollection 2019. PMID 30949343
- [Background] Neto T, Jacobsohn L, Carita AI, Oliveira R. Reliability of the Active-Knee-Extension and Straight-Leg-Raise Tests in Subjects With Flexibility Deficits. J Sport Rehabil. 2015 Dec 3;24(4):2014-0220. doi: 10.1123/jsr.2014-0220. Print 2015 Nov 1. PMID 25364856
- [Background] Khuman PR, Surbala L, Patel P, Chavda D. Immediate effects of single session post isometric relaxation muscle energy technique versus mulligan's bent leg raise technique on pain and hamstring flexibility in knee osteoarthritis participants: A randomised controlled study. Physiotherapy. 2014;3(9):324-35.
- [Background] Masekar MB, Rayjade DA, Yadav DT, Chotai DK. Effectiveness of Muscle Energy Technique and Proprioceptive Neuromuscular Facilitation in Knee Osteoarthritis.(2021). Int J Life SciPharmaRes.11(1):L16- 22.
- [Background] Marr M, Baker J, Lambon N, Perry J. The effects of the Bowen technique on hamstring flexibility over time: a randomised controlled trial. J Bodyw Mov Ther. 2011 Jul;15(3):281-90. doi: 10.1016/j.jbmt.2010.07.008. Epub 2010 Sep 15. PMID 21665103